CLINICAL TRIAL: NCT03444623
Title: Survivin as Predictive Biomarker for Development of Rheumatoid Arthritis
Brief Title: Survivin as Predictive Biomarker for RA
Acronym: SurviPred
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: Survivin rutin
Record Dates: First submitted 2018-02-05; First posted 2018-02-23 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Arthralgia; Joint Pain
Keywords: predictive factor; prognostic factor
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Purpose: to examine the possibility of using the onco-protein survivin as a predictive biomarker for identifying individuals at risk of developing rheumatoid arthritis within a cohort of patients seeking treatment for joint pain/stiffness. Secondly, to study survivin as a prognostic marker for joint destruction, refractory and highly active disease in patients with established RA.

DETAILED DESCRIPTION:
The study will analyse survivin levels in a non-selected material within a cohort of patients seeking help at their primary health care for joint pain, stiffness, swelling etc. Patients presenting with such symptoms (not explained by injury or other factors) are suspected to have an arthritic condition such as RA, and are routinely tested for presence of autoantibodies RF and ACPA. In this observational study we add measurement for survivin to the blood analyses of these patients. Information about patients expressing high levels of survivin will be reported to the referring doctor at the primary health care, and for patients not previously having been examined by a rheumatologist this will be offered.

The study will be performed at Sahlgrenska university hospital Gothenburg and Umeå university hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking treatment at the primary health care for problems with their joints (pain, stiffness).

Exclusion Criteria:

* Patients diagnosed with RA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seeking treatment at the primary health care for problems with their joints (pain, stiffness).
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Survivin positive | 1 year
  Survivin positive: > 0,45 ng/ml Survivin negative: < 0,45 ng/ml

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Rheumatology and Inflammation research, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erlandsson MC, Malmhall-Bah E, Chandrasekaran V, Andersson KME, Nilsson LM, Toyra Silfversward S, Pullerits R, Bokarewa MI. Insulin Sensitivity Controls Activity of Pathogenic CD4+ T Cells in Rheumatoid Arthritis. Cells. 2024 Dec 22;13(24):2124. doi: 10.3390/cells13242124. PMID 39768214